CLINICAL TRIAL: NCT06291844
Title: Ocular Trauma During the COVID-19 Pandemic Era at an Indonesian Tertiary Care Center: A Retrospective Cohort Study
Brief Title: Ocular Trauma and COVID-19 in Indonesia
Status: Completed | Type: Observational
Sponsor: Prof. R. D. Kandou General Hospital (Other)
Responsible Party: Principal Investigator, Vera Sumual, Vera Sumual, MD, PhD, Prof. R. D. Kandou General Hospital
Other Study IDs: Cohort-Mata-2023-1
Record Dates: First submitted 2024-03-01; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Ophthalmological Disorder; Ocular Injury; COVID-19
MeSH Terms: conditions — Eye Diseases; Eye Injuries; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ocular injuries, a significant contributor to avoidable blindness globally, impact approximately 55 million individuals each year. Prompt initial treatment is vital for improving vision, yet the scarcity of skilled eye specialists often results in overcrowding at advanced medical centers. Moreover, the COVID-19 outbreak has introduced distinct factors into the management of ocular trauma. This research investigated the epidemiology of ocular injuries during the pandemic and offered observations on the distinctive hurdles and trends encountered.

ELIGIBILITY:
Inclusion Criteria:

* Ocular Trauma Patients presenting between January 2021 to March 2022

Exclusion Criteria:

* Presenting on days outside the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ocular trauma patients
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Ocular Trauma | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Prof. R. D. Kandou General Hospital - Faculty of Medicine, Sam Ratulangi University, Manado, North Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No